CLINICAL TRIAL: NCT02400346
Title: Interventional, Open-label, Flexible-dose, Long-term Study to Evaluate the Safety and Tolerability of Brexpiprazole as Adjunctive Treatment in Elderly Patients With Major Depressive Disorder With an Inadequate Response to Antidepressant Treatment
Brief Title: Evaluation of the Safety of Adjunct Brexpiprazole in Elderly Patients With Major Depressive Disorder and an Inadequate Response to Antidepressant Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16160A; 2014-003547-35 (EudraCT Number)
Record Dates: First submitted 2015-03-17; First posted 2015-03-27 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-07

CONDITIONS: Major Depression Disorder

ARMS (1):
- Adjunct brexpiprazole (Experimental): All patients continue their current antidepressant treatment (ADT) and receive brexpiprazole in addition
  Interventions: Drug: Adjunct brexpiprazole; Drug: ADT

INTERVENTIONS:
Drug: Adjunct brexpiprazole — Weeks 1-4 titration from 0.5 up to 2 mg once daily, in weekly steps. For the rest of the 26 treatment weeks, maintenance with 1-3 mg once daily.
  Tablets for oral use once daily during 26 weeks. Tablet strengths: 0.5 mg, 1 mg, 2 mg and 3 mg.
Drug: ADT — Citalopram, ecitalopram, fluoxetine, sertraline, paroxetine IR, paroxetine CR, venlafaxine IR, venlafaxine XR (extended release), desvenlafaxine, duloxetine, mirtazapine, agomelatine, bupropion; dosing according to label

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of brexpiprazole as adjunctive treatment in an elderly population with major depressive disorder and an inadequate response to antidepressant treatment

ELIGIBILITY:
Main Inclusion Criteria:

* • The patient is a man or woman aged ≥65 yrs

  * The patient has Major Depressive Disorder according to Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM-IV-TR™).
  * The patient has an inadequate response to at least one adequate antidepressant treatment in the current Major Depressive Episode (MDE).
  * The patient has had the current MDE for ≥8 weeks
  * The patient is currently treated with a protocol specified ADT for at least 6 weeks
  * The patient is judged to benefit from adjunctive treatment with brexpiprazole according to the clinical opinion of the investigator.
  * Montgomery and Åsberg Depression Rating Scale (MADRS) total score > 18 at screening and baseline
  * Clinical Global Impression - Severity (CGI-S) total score ≥3 at screening and baseline

Main Exclusion Criteria:

* • The patient has a clinically significant unstable illness

  * The patient has newly diagnosed or unstable diabetes
  * The patient has a Mini Mental State Exam (MMSE) score <24
  * The patient has received Transcranial Magnetic Stimulation (TMS) and/or electroconvulsive therapy (ECT) less than 6 months prior to the Screening.
  * The patient, in the opinion of the investigator or based on Columbia-Suicide Severity Rating Scale (C-SSRS) Suicidal Ideation and behaviour rating, is at significant risk of suicide

Other protocol defined inclusion and exclusion criteria may apply

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 132 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (34):
- United States (13):
  - US012, Arcadia, California
  - US004, Miami, Florida
  - US007, Orlando, Florida
  - US006, Smyrna, Georgia
  - US002, O'Fallon, Missouri
  - US010, Toms River, New Jersey
  - US005, New York, New York
  - US008, New York, New York
  - US003, Staten Island, New York
  - US014, Oklahoma City, Oklahoma
  - US009, Allentown, Pennsylvania
  - US001, Memphis, Tennessee
  - US011, San Antonio, Texas
- Estonia (4):
  - EE002, Tallinn
  - EE001, Tartu
  - EE004, Tartu
  - EE003, Võru
- Finland (4):
  - FI001, Helsinki
  - FI002, Kuopio
  - FI003, Oulu
  - FI004, Tampere
- Germany (7):
  - DE002, Berlin
  - DE008, Berlin
  - DE003, Frankfurt
  - DE007, Hanover
  - DE006, Mittweida
  - DE001, Schwerin
  - DE005, Wiesbaden
- Poland (6):
  - PL006, Bialystok
  - PL003, Bydgoszcz
  - PL001, Chełmno
  - PL005, Gdansk
  - PL004, Lublin
  - PL002, Pruszcz Gdański

REFERENCES:
- [Derived] Lepola U, Hefting N, Zhang D, Hobart M. Adjunctive brexpiprazole for elderly patients with major depressive disorder: An open-label, long-term safety and tolerability study. Int J Geriatr Psychiatry. 2018 Oct;33(10):1403-1410. doi: 10.1002/gps.4952. Epub 2018 Jul 23. PMID 30039634

RESULTS

PARTICIPANT FLOW:
Groups:
- Adjunct Brexpiprazole: All patients continued their current antidepressant treatment and received brexpiprazole open-label in addition.
  Adjunct brexpiprazole administration was flexible and included a titration period: Weeks 1-4 titration from 0.5 up to 2 mg once daily, in weekly steps. For the rest of the 26 treatment weeks, maintenance with 1-3 mg once daily.
  Tablets for oral use once daily during 26 weeks. Tablet strengths: 0.5 mg, 1 mg, 2 mg and 3 mg.
Period: Overall Study
Arm/Group | Adjunct Brexpiprazole
Started | 132
Completed | 88
Not Completed | 44
Not completed — Adverse Event | 24
Not completed — Lack of Efficacy | 9
Not completed — Non-compliance with IMP | 1
Not completed — Withdrawal by Subject | 7
Not completed — Administrative or other reason(s) | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adjunct Brexpiprazole
Number analyzed (Participants) | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.4 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 130
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52
  Finland | 27
  Poland | 17
  Germany | 15
  Estonia | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment-Emergent Adverse Events
Description: Treatment-emergent adverse event is an adverse event that started or increased in intensity at or after baseline visit
Time Frame: Baseline to 30 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Adjunct Brexpiprazole
Number analyzed (Participants) | 132
Participants | 102

ADVERSE EVENTS:
Time Frame: Baseline to end of study (30 weeks)
Description: Treatment-Emergent Adverse Events are reported in this section
Arm/Group | Brex + ADT
All-Cause Mortality (participants affected / at risk) | 1/132
Serious Adverse Events (participants affected / at risk) | 6/132
Other Adverse Events (participants affected / at risk) | 79/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brex + ADT (N=132)
Acute myocardial infarction (Cardiac disorders) | 1
Myocardial rupture (Cardiac disorders) | 1
Postoperative wound infection (Infections and infestations) | 1
Eye contusion (Injury, poisoning and procedural complications) | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brex + ADT (N=132)
Fatigue (General disorders) | 20
Nasopharyngitis (Infections and infestations) | 8
Weight increased (Investigations) | 11
Increased appetite (Metabolism and nutrition disorders) | 13
Back pain (Musculoskeletal and connective tissue disorders) | 7
Akathisia (Nervous system disorders) | 11
Dizziness (Nervous system disorders) | 10
Headache (Nervous system disorders) | 7
Tremor (Nervous system disorders) | 9
Anxiety (Psychiatric disorders) | 10
Insomnia (Psychiatric disorders) | 8
Restlessness (Psychiatric disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No